CLINICAL TRIAL: NCT03438799
Title: A Multi-Center Observational Study to Collect Information Related to the Clinical Significance and Performance of the Cordio System
Brief Title: COMMUNITY STUDY- A Study to Collect Information for the Cordio System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cordio Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN 0011 (CLN0004, CA001); NCT03720509 (obsolete NCT alias); NCT03720535 (obsolete NCT alias)
Record Dates: First submitted 2018-02-11; First posted 2018-02-20 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cordio: Cordio R&D database to develop the Cordio System
  Interventions: Device: Cordio System

INTERVENTIONS:
Device: Cordio System — App, cloud and web device

SUMMARY:
This is a multi-center, observational, non-interventional, prospective, Single-arm, open study for database establishment for R&D purposes. R&D data will be analyzed retrospectively in order to validate algorithm efficacy.

The study will be conducted in the following settings: outpatinets clinics

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Symptomatic Heart Failure Patient.
3. The patient is willing to participate as evidenced by signing the written informed consent.
4. Male or non-pregnant female patient.

Exclusion Criteria:

1. Subject who, in the Investigator's opinion, unable to comply with the daily use of the App due to mental disorders (e.g., depression, dementia).
2. Patient who has had a major cardiovascular event (e.g., myocardial infraction, stroke) within 3 months prior to screening visit.
3. Patient with severe alcohol or drug use.
4. Psychological instability, inappropriate attitude or motivation.
5. Patient with life threatening debilitating disease other than cardiac.
6. Subject currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NYHA 2-3. All patients must meet eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-10-20 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
R&D Database & Efficiency | 2 years
  Building R&D recording database and retrospectively Cordio System needs to reach correlation between the system generated alerts to HF exacerbation

SECONDARY OUTCOMES:
Usability | 2 years
  Questionnaires with SUS scale and specific app questions in order to assess the app usability

OTHER OUTCOMES:
SADE Endpoint | 2 years
  Demonstration of the safe use of the device by overall incidence of device related adverse events.

CONTACTS AND LOCATIONS:
Locations (8):
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Clalit Bat Yam, Bat Yam
  - Clalit Be'er Sheva, Beersheba
  - Clalit Bet Shemesh, Bet Shemesh
  - Shamir Medical Center, Be’er Ya‘aqov
  - Hillel Yaffe Medical Center, Hadera
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No